CLINICAL TRIAL: NCT02897635
Title: Developing an Integrative Ayurvedic Intervention for Breast Cancer Survivorship
Brief Title: Integrative Approaches For Cancer Survivorship 2: Project 1
Acronym: IACS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-18567
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Integrative Medicine Intervention (Experimental): Study participants will attend 14 visits with an integrative medicine clinician over the course of 6 months followed by a 6 month maintenance phase. The treatment modalities employed in the study will include nutrition and lifestyle recommendations.
  Interventions: Behavioral: Individualized Integrative Medicine Intervention

INTERVENTIONS:
Behavioral: Individualized Integrative Medicine Intervention

SUMMARY:
The purpose of this study is to develop and test a 12-month Integrative Medicine intervention based on Ayurvedic medicine in recent breast cancer survivors.

DETAILED DESCRIPTION:
Cancer associated symptoms and impaired quality of life remain significant problems for patients despite advances in cancer treatment. Few effective treatment options exist for these symptoms. Integrative medicine is rising in popularity in the United States; however, few integrative medicine modalities have been rigorously studied. Ayurveda, a whole system of medicine that originated in the Indian subcontinent, has its own system of diagnostics and therapeutics, and among its strengths are wellness and prevention. The investigators aim to perform a prospective single arm clinical study of a manualized Ayurvedic approach in breast cancer survivors with impaired quality of life. Specifically, the investigators aim to refine the manualized Ayurvedic intervention; to assess feasibility; and to determine whether clinically meaningful effects can be achieved with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer survivor who is over 1 month and less than 24 months beyond the completion of primary therapy (surgery, radiation, and chemotherapy)
* Having received chemotherapy as part of their primary therapy for breast cancer
* Be in complete remission
* Aged 18 years or older
* Able to read, write, and understand English
* Karnofsky Performance Status (KPS) greater than or equal to 60
* Have impaired quality of life
* Ability to give informed consent

Exclusion Criteria:

* Having received Ayurvedic treatment within 6 months of study enrollment
* Receiving chemotherapy or radiotherapy at the time of study enrollment. Anti-her2 directed therapy is not exclusionary.
* Being within 1 month (before or after) of surgery for breast cancer (including breast reconstructive surgery). Smaller surgical procedures such as implant exchange are not exclusionary.
* Patients on adjuvant hormone therapy for less than 2 months
* Have surgery for breast cancer or breast reconstructive surgery planned during the initial 6 month study period. Smaller surgical procedures such as implant exchange are not exclusionary.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Change in quality of life over 12 months | Baseline, 3 months, 6 months, 12 months
  The investigators will use the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30) in conjunction with a Breast Cancer-Specific Subscale (BR23) to collect data on qualify of life and cancer-related symptoms.

SECONDARY OUTCOMES:
Change in fatigue over 12 months | Baseline, 3 months, 6 months, 12 months
  The investigators will use the Lee Fatigue Scale (LFS) to collect data on fatigue.
Change in sleep quality over 12 months | Baseline, 3 months, 6 months, 12 months
  The investigators will use the General Sleep Disturbance Scale (GSDS) to collect data on sleep disturbance.
Change in anxiety over 12 months | Baseline, 3 months, 6 months, 12 months
  The investigators will use the Spielberger State Anxiety Inventory (STAI-S) to collect data on anxiety.
Change in depressive symptoms over 12 months | Baseline, 3 months, 6 months, 12 months
  The investigators will use the Center for Epidemiological Studies - Depression Scale (CES-D) to collect data on depressive symptoms.
Change in pain over 12 months | Baseline, 3 months, 6 months, 12 months
  The investigators will use the Brief Pain Inventory (BPI) to collect data on pain intensity and interference with function.
Change in diet over 12 months | Baseline, 3 months, 6 months, 12 months
  The investigators will use the Automated Self-Administered 24-hour Recall (ASA24) to assess dietary recall over a 24 hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Dhruva, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Osher Center for Integrative Medicine, San Francisco, California, United States